CLINICAL TRIAL: NCT06814418
Title: The Effect of Injectable Platelet Rich Fibrin (iPRF) in Non-surgical Periodontal Treatment- A Randomized Controlled Clinical Trial
Brief Title: Injectable Platelet Rich Fibrin in Periodontal Treatment
Acronym: I-PRF
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Aristotle University Of Thessaloniki (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 234/21-03-2023
Record Dates: First submitted 2024-11-27; First posted 2025-02-07 (Actual); Last update posted 2025-02-07 (Actual); Status verified 2025-01

CONDITIONS: Periodontitis
Keywords: Periodontitis; Platelet Rich Fibrin; Non surgical; Porphyromonas gingivalis; Filifactor alocis; Pocket closure
MeSH Terms: conditions — Periodontitis | interventions — proliferation regulatory factors, human urine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Test (Experimental): Non-surgical periodontal treatment + injectable Platelet Rich Fibrin
  Interventions: Procedure: Non-surgical periodontal treatment; Procedure: Injectable Platelet Rich Fibrin (I-PRF)
- Control (Active Comparator): Non-surgical periodontal treatment
  Interventions: Procedure: Non-surgical periodontal treatment

INTERVENTIONS:
Procedure: Non-surgical periodontal treatment — Step I and II of periodontal treatment.
Procedure: Injectable Platelet Rich Fibrin (I-PRF) — Infusion of I-PRF in sited with PPD≥5mm.
  Arms: Test

SUMMARY:
The aim of this randomized controlled parallel clinical trial is to investigate the efficacy of injectable Platelet Rich Fibrin (iPRF) as an adjunctive to non-surgical periodontal therapy (STEP 1 & 2 of periodontal treatment).

Thirty-two (32) patients diagnosed with stage III periodontitis will be randomly assigned to two study groups. Participants will receive non-surgical periodontal treatment only (control group) or non-surgical periodontal treatment with iPRF (test group). Patients will receive step 1 and 2 of periodontal treatment. Step 2 of periodontal treatment will be completed in one visit. Test group also will receive immediately after the subgingival instrumentation iPRF at the sites with PPD≥5mm.

Subgingival plaque will be collected with paper points at different time points- baseline: before treatment, 3 and 6 months after treatment.

The presence and quantification of bacteria: -Porphyromonas gingivalis (Pg), Filifactor Alocis (F.Alocis)- will be examined with quantitative polymerase chain reaction (q PCR). Clinical parameters, including bleeding on probing (BOP), probing pocket depth (PPD), clinical attachment level (CAL), gingival recession (REC) will be recorded at baseline, 3 and 6 months after treatment.

Patient satisfaction will be assessed through questionnaires regarding quality of life, pain perception and the use of analgesics. The questionnaires will be completed one week after subgingival instrumentation.

ELIGIBILITY:
Inclusion Criteria:

* Ages Eligible for Study: >18 years old (Adults)
* Diagnosed Periodontitis Stage III
* Presence of ≥ 15 teeth
* Signed written consent form by patient

Exclusion Criteria:

* At least one edentulous jaw
* Need for chemoprophylaxis before treatment
* Periodontal treatment the last 6 months
* Antibiotic treatment the last 6 months
* Immunomodulatory diseases (e.g. diabetes mellitus, rheumatoid arthritis, osteoporosis), for which patients do not take medication
* HbA1c> 7.0% in patients with diabetes
* Pregnancy/ Lactation
* Medications or undergoing treatment which may affect mucosal healing

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Estimated)
Dates: Start 2023-06-15 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-10 (Estimated)

PRIMARY OUTCOMES:
Pocket closure - Percentage of successful treatment outcome | 6 months
  Pocket closure : clinical Periodontal Marker: probing pocket depth (PPD) ≤4 mm and absence of bleeding on probing (BOP). (Periodontal probe UNC15, Hu-Friedy, Rotterdam, the Netherlands)
Bleeding on Probing (BoP) - Change in percentage | 6 months
  Clinical Periodontal Marker: Bleeding after slight pressure by a standardized (dimensions and shape) periodontal probe with a controlled (∼0.25 N) force to the apical end of the sulcus (Periodontal probe UNC15, Hu-Friedy, Rotterdam, the Netherlands)
Clinical Attachment Loss (CAL) | 6 months
  Clinical Periodontal Marker: The distance in mm from the CEJ to the gingival margin (Periodontal probe UNC15, Hu-Friedy, Rotterdam, the Netherlands)

SECONDARY OUTCOMES:
Microbiological Assessment | 6 months
  Presence and quantification of bacteria: -Porphyromonas gingivalis (Pg), Filifactor Alocis (F.Alocis)- will be examined by quantitative polymerase chain reaction (qPCR).
  Reduction or absence of these specific bacteria leads to reduction of inflammation and results in non-progression of periodontal disease (reduction of probing depth (PPD), gain of clinical attachment level (CAL), less bleeding on probing (BOP) and pocket closure )
Patient-reported Outcomes | 1 week
  Patient-reported outcomes will be assessed using the McGill Pain Questionnaire-2 (SF-MPQ-2) short form.
  It includes 22 descriptors, each descriptor is rated on a 0-10 numerical scale, where 0 = no pain and 10 = worst possible pain, reflecting the severity of each pain characteristic over the past week.
Analgesic Intake | 1 week
  The number and type of analgesics taken by the patient will be recorded for each individual day during the week following the treatment

CONTACTS AND LOCATIONS:
Overall Officials: Leonidas Batas, Ass. Professor, DDS, MSc, PhD, Study Director — Aristotle University Of Thessaloniki; Sofia Zarenti, DDS, Principal Investigator — Aristotle University Of Thessaloniki
Locations (1):
- Aristotle University of Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Ferrarotti F, Baima G, Rendinelli M, Citterio F, Mariani GM, Mussano F, Romano F, Romandini M, Aimetti M. Pocket closure after repeated subgingival instrumentation: a stress test to the EFP guideline for stage III-IV periodontitis. Clin Oral Investig. 2023 Nov;27(11):6701-6708. doi: 10.1007/s00784-023-05279-6. Epub 2023 Sep 29. PMID 37773418
- [Background] D'Aiuto F, Ready D, Parkar M, Tonetti MS. Relative contribution of patient-, tooth-, and site-associated variability on the clinical outcomes of subgingival debridement. I. Probing depths. J Periodontol. 2005 Mar;76(3):398-405. doi: 10.1902/jop.2005.76.3.398. PMID 15857074
- [Background] Moraschini V, Miron RJ, Mourao CFAB, Louro RS, Sculean A, da Fonseca LAM, Calasans Maia MD, Shibli JA. Antimicrobial effect of platelet-rich fibrin: A systematic review of in vitro evidence-based studies. Periodontol 2000. 2024 Feb;94(1):131-142. doi: 10.1111/prd.12529. Epub 2023 Sep 22. PMID 37740425
- [Background] Ozcan E, Saygun I, Kantarci A, Ozarslanturk S, Serdar MA, Ozgurtas T. The effects of a novel non-invasive application of platelet-rich fibrin on periodontal clinical parameters and gingival crevicular fluid transforming growth factor-beta and collagen-1 levels: A randomized, controlled, clinical study. J Periodontol. 2021 Sep;92(9):1252-1261. doi: 10.1002/JPER.20-0713. Epub 2021 Jan 15. PMID 33382101
- [Background] Narendran N, Anegundi RV, Shenoy SB, Chandran T. Autologous platelet-rich fibrin as an adjunct to non-surgical periodontal therapy-A follow up clinical pilot study. Wound Repair Regen. 2022 Jan;30(1):140-145. doi: 10.1111/wrr.12979. Epub 2021 Oct 22. PMID 34687113
- [Background] Al-Rihaymee S, Sh Mahmood M. The efficacy of non-surgical platelet-rich fibrin application on clinical periodontal parameters and periostin level in periodontitis: Clinical trial. J Cell Mol Med. 2023 Feb;27(4):529-537. doi: 10.1111/jcmm.17675. Epub 2023 Jan 23. PMID 36691719
- [Background] Sharma A, Pradeep AR. Autologous platelet-rich fibrin in the treatment of mandibular degree II furcation defects: a randomized clinical trial. J Periodontol. 2011 Oct;82(10):1396-403. doi: 10.1902/jop.2011.100731. Epub 2011 Feb 2. PMID 21284545
- [Background] Bajaj P, Pradeep AR, Agarwal E, Rao NS, Naik SB, Priyanka N, Kalra N. Comparative evaluation of autologous platelet-rich fibrin and platelet-rich plasma in the treatment of mandibular degree II furcation defects: a randomized controlled clinical trial. J Periodontal Res. 2013 Oct;48(5):573-81. doi: 10.1111/jre.12040. Epub 2013 Jan 14. PMID 23317096
- [Background] Ajwani H, Shetty S, Gopalakrishnan D, Kathariya R, Kulloli A, Dolas RS, Pradeep AR. Comparative evaluation of platelet-rich fibrin biomaterial and open flap debridement in the treatment of two and three wall intrabony defects. J Int Oral Health. 2015 Apr;7(4):32-7. PMID 25954068
- [Background] Thorat M, Pradeep AR, Pallavi B. Clinical effect of autologous platelet-rich fibrin in the treatment of intra-bony defects: a controlled clinical trial. J Clin Periodontol. 2011 Oct;38(10):925-32. doi: 10.1111/j.1600-051X.2011.01760.x. Epub 2011 Jul 21. PMID 21777267
- [Background] Pradeep AR, Rao NS, Agarwal E, Bajaj P, Kumari M, Naik SB. Comparative evaluation of autologous platelet-rich fibrin and platelet-rich plasma in the treatment of 3-wall intrabony defects in chronic periodontitis: a randomized controlled clinical trial. J Periodontol. 2012 Dec;83(12):1499-507. doi: 10.1902/jop.2012.110705. Epub 2012 Feb 21. PMID 22348695
- [Background] Sharma A, Pradeep AR. Treatment of 3-wall intrabony defects in patients with chronic periodontitis with autologous platelet-rich fibrin: a randomized controlled clinical trial. J Periodontol. 2011 Dec;82(12):1705-12. doi: 10.1902/jop.2011.110075. Epub 2011 Apr 5. PMID 21513477
- [Background] Miron RJ, Zucchelli G, Pikos MA, Salama M, Lee S, Guillemette V, Fujioka-Kobayashi M, Bishara M, Zhang Y, Wang HL, Chandad F, Nacopoulos C, Simonpieri A, Aalam AA, Felice P, Sammartino G, Ghanaati S, Hernandez MA, Choukroun J. Use of platelet-rich fibrin in regenerative dentistry: a systematic review. Clin Oral Investig. 2017 Jul;21(6):1913-1927. doi: 10.1007/s00784-017-2133-z. Epub 2017 May 27. PMID 28551729